CLINICAL TRIAL: NCT03887611
Title: A Multi-center Study of Differential Diagnosis Thyroid Nodules by Ultrasound Artificial Intelligence and Ultrasound Elastography
Brief Title: Application of Ultrasound Artificial Intelligence and Elastography in Differential Diagnosis of Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xin-Wu Cui (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Macheng People's Hospital (Unknown); Huangshi Central Hospital (Other); Affiliated Hospital of Jiangsu University (Other); The First People's Hospital of Yichang (Unknown); Yichang Second People's Hospital (Other); Xiangyang Central Hospital (Other); The Second Hospital of Anhui Medical University (Other); Anqing People's Hospital (Unknown); Huainan People's Hospital (Unknown); Taizhou Hospital (Other); Wenzhou Central Hospital (Other); Xuzhou First People's Hospital (Unknown); The Central Hospital of Lishui City (Other); Huai'an First People's Hospital (Other); WISCO General Hospital (Unknown); Jiangxia District First People's Hospital (Unknown); Enshi State Central Hospital (Unknown); Lianyungang Third People's Hospital (Unknown); First People's Hospital of Xianyang (Other)
Responsible Party: Sponsor-Investigator, Xin-Wu Cui, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 2019(S074)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Thyroid Nodule
Keywords: Artificial Intelligence; Ultrasound;Thyroid nodule; ECI
MeSH Terms: conditions — Thyroid Nodule | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- thyroid nodules: Those with one or more breast nodules, age 18 or older, upcoming FNAB or surgery and signed informed consent.Those without adverse effects on the test or threatening other candidates, such as mental illness, pregnancy, poor ultrasound image quality, history of thyroid surgery or thyroid biopsy, simple cystic nodules, calcification, excessive mass or too small, the S-DetectTM system can not identify the boundary of the tumor, the basic information is incomplete.
  Interventions: Device: Ultrasound diagnosis

INTERVENTIONS:
Device: Ultrasound diagnosis — Ultrasound diagnosis of lesions with Samsung S-Detect and ECI technology

SUMMARY:
The application of computer-aided diagnosis (CAD) technology "S-DetectTM" enables qualitative and quantitative automated analysis of ultrasound images to obtain objective, repeatable and more accurate diagnostic results. The Elastic Contrast Factor (ECI) technique, unlike conventional strain-elastic imaging techniques, can evaluate the elastic distribution in the region of interest. The purpose of the study was to evaluate the differential diagnosis value of ultrasound S-DetectTM technology for benign and malignant thyroid nodules and evaluate the consistency of ultrasound S-DetectTM technology and sonographer in the differential diagnosis of thyroid nodules and explore the differential diagnosis value of Samsung ultrasound ECI technology for benign and malignant thyroid nodules.

DETAILED DESCRIPTION:
Thyroid nodules are one of the most common nodular lesions in adults, and their incidence is increasing. Clinical studies have found that about 10%-15% of adults have thyroid nodules, most of which are benign nodules, only 7% of thyroid nodules tend to be malignant, but if not treated promptly, 5% of patients will still from benign to malignant. The incidence of thyroid cancer increases with age. According to the National Cancer Research Center, about 64,300 new cases of thyroid cancer occurred in the world in 2016, and about 1,980 died of thyroid cancer. Timely and accurate detection of thyroid nodules and differentiation of benign and malignant are important for improving clinical treatment and improving patient prognosis.

S-Detect technology is a computer-aided (CAD) system recently developed by Samsung Medical Center for thyroid ultrasound to assist in morphological analysis based on the Thyroid Imaging Reporting and Data System (TI-RADS) description and final assessment.This provides a new way to identify the benign and malignant thyroid nodules.

The ECI technique, unlike conventional strain-elastic imaging technology, performs an elastic analysis of the entire two-dimensional image. Moreover, when measuring the elastic ratio, it is only necessary to place a region of interest (ROI) at the nodule. Compared with the average elasticity of the surrounding area, it is more reflective of the elastic ratio of the mass to the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Had thyroid lesions detected by ultrasound
2. Age 18 or older
3. Upcoming FNAB or surgery
4. Signing informed consent

Exclusion Criteria:

1. Patients who had received a biopsy of thyroid lesion before the ultrasound examination
2. Can not cooperate with the test operation
3. Patients who were pregnant or lactating
4. Patients who were undergoing neoadjuvant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid nodules in large tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-01-18 (Estimated); Study Completion 2020-03-18 (Estimated)

PRIMARY OUTCOMES:
Benign or malignant lesions as determined by pathology | Before surgery or biopsy
  The pathological diagnosis of benign or malignant lesions from surgery samples
Elastic ratio | Before surgery or biopsy
  Clear ECI value

CONTACTS AND LOCATIONS:
Overall Officials: Xin-Wu Cui, PhD,MD, Study Chair — Tongji Hospital; You-Bin Deng, PhD,MD, Study Chair — Tongji Hospital
Locations (1):
- Xin-Wu Cui, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not public because of the personal information of the participants

REFERENCES:
- [Result] Choi YJ, Baek JH, Park HS, Shim WH, Kim TY, Shong YK, Lee JH. A Computer-Aided Diagnosis System Using Artificial Intelligence for the Diagnosis and Characterization of Thyroid Nodules on Ultrasound: Initial Clinical Assessment. Thyroid. 2017 Apr;27(4):546-552. doi: 10.1089/thy.2016.0372. Epub 2017 Feb 28. PMID 28071987